CLINICAL TRIAL: NCT05813821
Title: Evaluation of a National Antibiotic Stewardship Intervention (7-VINCut) to Decrease the Duration of Antibiotic Treatment and Carbapenem Use in Surgical Services
Brief Title: 7-VINCut Antibiotic Stewardship Intervention to Decrease Duration of Antibiotic Treatment and Carbapenem Use in Surgery
Acronym: 7_VINCUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep Maria Badia, Prof, Hospital de Granollers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HGG2022_01
Record Dates: First submitted 2023-03-30; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Medication Adherence; Antibiotic Resistance, Microbial; Medication Errors and Other Product Use Errors and Issues
Keywords: Anti-Bacterial Agents / therapeutic use; Infection Control / organization & administration; Antimicrobial Stewardship / organization & administration; Antimicrobial Stewardship / statistics & numerical data; General Surgery / standards
MeSH Terms: conditions — Medication Adherence | interventions — Antimicrobial Stewardship; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, interventional, cohort study analysing the effect of an antimicrobial stewardship intervention in surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with antibiotic treatment in surgical departments (Experimental): All patients admitted for antibiotic treatment in the surgical departments of the participating centres were included.
  Interventions: Behavioral: Antimicrobial stewardship in surgery

INTERVENTIONS:
Behavioral: Antimicrobial stewardship in surgery — Hospitals were invited to form a surgical antibiotic stewardship program (ASP) with surgeons, pharmacists and infectious disease specialists. The interventional ASP relied on an audit and feedback strategy to issue recommendations aimed at reducing the duration of antibiotic treatment and the use of drugs with a particular impact on microbial ecology.
  All patients hospitalized in surgical departments were prospectively analyzed weekly. A computerized alert allowed the ASP team to identify patients with antibiotic treatment >7 days. The team meet to discuss the appropriateness of each antibiotic treatment, issuing a written recommendation for each patient. The intervention was performed only once for each patient, except if they had a new focus of infection. The recommendations available for prolonged treatments were: withdraw, maintain, de-escalate, broaden, change route, optimize dose, no recommendation. Adherence to the recommendations was recorded 48 hours later by the ASP team.

SUMMARY:
Antimicrobial resistance (AMR) is one of the top ten public health threats facing humanity. The misuse and overuse of antibiotics has been identified as a major factor in the development of drug-resistant pathogens, and 30% of all antimicrobials administered in Western acute hospitals are unnecessary or inappropriate. As a consequence, the establishment of antimicrobial stewardship programmes (ASPs) has increased in hospitals over the past decades.

Using ASPs to optimise antimicrobial use is critical to effectively fight infections, protect patients and reduce AMR. ASPs can increase infection cure rates while reducing AMR, but it has been reported that few of them are specifically targeted at surgical specialties or led by surgeons.

Surgeons are actively involved in antibiotic prescribing and should therefore play an important role in the development and leadership of ASPs in surgical departments.

Practice Guidelines have established recommendations for the wise use of antibiotics in patients affected by intra-abdominal infection: early identification of sepsis, early initiation of antimicrobial therapy and early control of the infectious focus. The literature on the optimal duration of antibiotic treatment in surgery is sparse, but it seems that, if the septic source has been effectively controlled, short courses of treatment show the same results as longer courses.Compliance rates with the suggested duration of treatment in evidence-based guidelines are low among the surgical community.

No specially designed ASPs for the reduction of treatment duration in surgery have been reported. ASPs may be easy to introduce in a single hospital, but the feasibility of a nationwide implementation of ASPs in a large and diverse hospital population is unclear.

This prospective, interventional, cohort study was aimed: to reduce the duration of antimicrobial treatment in surgical departments by modifying their prescriptions through educational and consensual interventions; and to assess the feasibility of implementing a multi-centre ASP, leveraging a nationwide surveillance programme for healthcare-associated infection.

It was hypothesised that a coordinated and guided implementation strategy, organised within a consolidated infection surveillance network, would lead to the successful implementation of the ASP and reduce antibiotic consumption in participating hospitals.

DETAILED DESCRIPTION:
This is a multicenter, prospective, interventional, cohort study analysing the effect of an antimicrobial stewardship intervention in surgery. The study uses data collected prospectively leveraging an infection surveillance network.

4.1. Setting and patients. The 7VINCut antibiotic stewardship program started in 2019 at national level to shorten the duration of antibiotic therapy in adult patients admitted to surgical departments. Secondary objectives were to reduce the consumption of carbapenems in surgical services and to reduce the consumption of other antibiotics with ecological impact (piperacillin-tazobactam, amoxicillin/clavulanate, 3rd and 4th generation cephalosporins and quinolones).

The prospective study was conducted between January 2019 and December 2022. Data from 32 hospitals participating in the network were included in the analysis.

All patients aged 18 years or older admitted to general and urological surgical services, who received systemic antibiotic treatments lasting for 7 or more days were included. Patients with antibiotics prescribed for surgical prophylaxis were excluded. Because to the characteristics of the infections treated in Orthopedics and Vascular Surgery departments, often requiring long-term treatments, the cases with diseases specific to these services (osteomyelitis, diabetic foot, etc) were excluded.

4.2. Intervention. The intervention started with the dissemination of the project protocol to all hospitals participating in the network, and a workshop for surgical and infection control teams. This was a multidisciplinary project in which hospitals were invited to form a specific surgical ASP with surgeons, pharmacists and infectious disease specialists. Participating institutions established local teams with the support of senior hospital leaders to facilitate the implementation of the ASP.

The interventional ASP relied on an audit and feedback strategy to issue recommendations aimed at reducing the duration of antibiotic treatment regimens and reducing the use of drugs with a particular impact on microbial ecology.

All patients hospitalized in the targeted departments were prospectively analyzed weekly. A computerized alert allowed the ASP team to identify those patients whose antibiotic treatment lasted longer than 7 days. The team meet to discuss the appropriateness of each antibiotic treatment, issuing a written recommendation for each patient. The intervention was performed only once for each patient, except if they had a new focus of infection. The recommendations available for prolonged treatments were: withdraw, maintain, de-escalate, broaden, change route, optimize dose, no recommendation. The recommendations were discussed in the Surgery Departments and implemented if deemed necessary. Adherence to the recommendations was recorded 48 hours later by the ASP team.

Although the intervention focused on the duration of antibiotic treatment, the stewardship team added recommendations on the microbiological appropriateness of the treatments and the use of broad-spectrum antibiotics, especially carbapenems. Before implementation of the program in the hospital, a series of educational initiatives related to antibiotic management in the Department of Surgery were introduced.

The prescriptions analyzed were either pathogen directed or empirical broad spectrum antibiotic treatments. Before making the ASP recommendations, the microbiological results were reviewed, when available. The appropriateness of the empirical antibiotics prescribed according to the hospital antibiotic guideline was also reviewed.

The main outcome evaluated was the percentage of patients subjected to more than 7 days of antibiotic therapy. Other outcomes were: percentage of new patients on antibiotic treatment >7 days out of the total number of patients on antibiotic treatment admitted to the surgical services; percentage of adherence to recommendations.

Variables such as type of infection, quality of control of infectious focus (good, uncertain, bad) for which antibiotic treatment was indicated was reported, use of broad spectrum antibiotics, route of administration, and microbiological adequacy have been analyzed.

4.3. Ethics and statistics. The study was approved by the Research Ethics Committee of the Hospital General Universitari de Granollers with code 20222042, which did not consider an informed consent document necessary. The project will be reported according to the "Strengthening the reporting of cohort, cross-sectional and case-control studies in surgery" (STROCSS 2021) criteria.

Data was entered into a computerized database that was analyzed using the IBM SPSS program (v. 21.0, Chicago, IL, USA). The evolution of the percentage of new patients undergoing a prolonged antibiotic treatment related to the total number of patients on antibiotic treatment has been evaluated by simple linear regression. The linear relationship was tested by ANOVA tests and Pearson's correlation coefficients (Pc) were obtained. Values of p ≤ 0.05 were considered statistically significant. A bilateral distribution was assumed for all p values.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the targeted surgical departments

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32499 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patients subjected to more than 7 days of antibiotic therapy | One week
  Percentage of patients subjected to more than 7 days of antibiotic therapy in surgical departments

SECONDARY OUTCOMES:
Compliance with recommendations issued by stewardship teams | 2 days after recommendation
  The number of patients in which the recommendations of the ASP team have been followed will be analysed out of the total number of recommendations issued. This will be done by reviewing electronic medical records and calculating the percentage of compliance with the recommendations out of the total number of antibiotic treatment recommendations issued by the management team.
Type of infection | One week
  Type of infection for which antibiotic treatment was indicated
Quality of control of septic focus | Two days
  The assessment team will analyse the quality of focus control for each case, looking at the surgeon's subjective assessment at the end of the operation (recorded in the operative notes) and the clinical evolution of the patient during the first two days post-operatively. Quality shall be classified as good, uncertain or poor.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Badia, Study Director — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain